CLINICAL TRIAL: NCT03827577
Title: OMEGA, A Randomized Trial of Local Ablative Therapy Vs. Conventional Treatment in Oligometastatic NSCLC
Brief Title: OMEGA, Local Ablative Therapy in Oligometastatic NSCLC
Acronym: OMEGA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other); San Luigi Gonzaga Hospital (Other); Regina Elena Cancer Institute (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Azienda Ospedaliera San Camillo Forlanini (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1533CESC
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAT arm (Experimental): Lung resection (if primary in place) + local ablative therapy of all metastatic sites + standard medical treatment.
  patients may be enrolled either before any systemic therapy or after 3 months of treatment without progression according to local coordinator decision
  Interventions: Procedure: Surgical removal of primary and/or of all oligometastases; Radiation: Non-surgical LAT; Drug: Standard medical therapy
- Control Arm (Active Comparator): Standard medical treatment
  Local ablative therapy on the brain will be administered in any case to patients harboring cerebral oligometastases
  Interventions: Drug: Standard medical therapy

INTERVENTIONS:
Procedure: Surgical removal of primary and/or of all oligometastases — Standard lobectomy or segmentectomy if tumor resectable without pneumonectomy (prefer lobectomy if cardiorespiratory function is not or only moderately compromised, prefer segmentectomy if primary tumor less than 2 cm or cardiorespiratory function is more than moderately compromised but still permissive) Mediastinal lymph node dissection (at least 8 lymphnodes from at least 3 stations including station 7).
  Arms: LAT arm
Radiation: Non-surgical LAT — Non-surgical LAT may be carried out either by SABR or SBRT or RFA according to site of metastasis, local expertise and availability of resources.
  Arms: LAT arm
Drug: Standard medical therapy — platinum-based doublet according to local protocols or targeted agents according to EGFR/ALK/ROS-1 mutational status or immunotherapy agents according to PDL1 expression.

SUMMARY:
Oligometastatic lung cancer (OM-NSCLC) seems to be associated with a better prognosis than usual Stage IV non-small cell lung cancer when radical local therapy of all metastatic sites is administered but the impact of such an approach on overall survival and quality of life remains to be defined by adequately powered phase III trials.

A consortium of tertiary referral centres involved in Lung Cancer management at the national level was established to launch a randomized trial of local ablative therapy in OM-NSCLC patients with potentially resectable or locally controlled primary tumors has been designed.

Inclusion criteria include adequate performance status, primary tumor controlled or controllable staging with whole-body FDG PET scan and brain MRI, fit to receive at least 3 cycles of platinum-based doublet chemotherapy, or immunotherapy or targeted agents according to molecular profile.

Exclusion criteria include cerebral oligometastasis alone (will receive local therapy in any case), metastasis in sites where normal radiotherapy constraints cannot be met, multiple subsolid nodules in the absence of extrapulmonary metastasis, prior malignant tumor with some exceptions, relevant co-morbidities that would significantly reduce life expectancy on their own.

Patients with synchronous or metachronous oligometastatic lung cancer (1-3 metastatic lesions) will be randomized to local ablative therapy + standard treatment Vs. standard treatment. Balancing between study arms will be performed according to synchronous vs. metachronous presentation, Number of oligometastases, Nodal status and Oncogene-addiction or PDL-1 expression. Primary outcome will be Overall Survival (OS) from randomization. The sample size is set to 195 patients.

Disease state and life status will be assessed on a 3-monthly basis by physical examination, whole-body CT scan plus repeat PET-scan if needed and Brain MRI if brain metastasis at enrolment. Toxicity and adverse events will be assessed according to NCI-Common Terminology Criteria. And RTOG criteria. Quality of life will be assessed at randomization and after six months by the SF36/LCSS

DETAILED DESCRIPTION:
Lung cancer is a systemic disease with local manifestations that are ultimately responsible for a reduced life expectancy in a relatively large subgroup of metastatic lung cancer patients.

In such a subgroup, local ablative therapy of the primary tumor and of all metastatic lesions with a combination of surgery and/or radiotherapy should lead to a clinically significant improvement of their overall survival with acceptable morbidity and preserved Quality of Life compared with medical treatment alone

OMEGA is a randomized trial of local ablative therapy in NSCLC patients with potentially resectable or locally controlled primary tumors and oligometastatic disease

The decision to randomise OM-NSCLC patients either before any systemic therapy or after 3 months of treatment without progression is left to the recruiting centre(s).

Local ablative therapy will be administered in any case to patients harboring cerebral oligometastasis

Statistical methods

Dynamic balancing as per the method of Pocock and Simon [16] according to:

* Synchronous vs. metachronous presentation
* Number of oligometastases (1 vs. 2-3) including extrathoracic N3 disease
* Nodal status (N0 vs. N+)
* Oncogene-addiction (EGFR/ALK/ROS-1 driven or PDL1 >50% vs <50% vs. wild type)

ELIGIBILITY:
Inclusion criteria

* ECOG performance status 0-1 at the time of randomization
* Pathologically confirmed NSCLC.
* Staging with whole-body FDG PET scan and brain MRI or CT with IV contrast.
* Between 1 and 3 metastatic lesions, assessable according to RECIST v1.1 and suitable for LAT prior to trial registration.
* Primary tumor controlled (metachronous oligometastasis) or resectable/suitable for ablative radiotherapy.
* Patient is deemed fit to receive at least 3 cycles of platinum-based doublet chemotherapy, cisplatin or carboplatin, according to local guidelines.
* If pulmonary involvement, it must be bilateral with at least 3 lung lesions, or extrapulmonary metastasis must be present
* If brain involvement, up to 2 brain metastases, the largest brain lesion < 3cm in maximum diameter at the time of randomization.

Exclusion criteria

* Any tumor site besides brain metastasis requiring immediate LAT for palliation.
* Patient has received previous LAT for extra-cerebral metastasis
* Patient has received previous systemic treatment for his/her NSCLC malignancy and is experiencing disease progression at the time of randomization (except adjuvant chemotherapy and/or radiotherapy more than 6 months earlier)
* Patient has had palliative radiotherapy to any tumor site prior to registration and/or requires palliative radiotherapy prior to randomization.
* High clinical suspicion of direct invasion of the wall of any major blood vessel or medulla by the primary tumor or metastasis
* Brain metastasis within the brainstem, or leptomeningeal disease.
* Metastasis in sites where normal radiotherapy constraints cannot be met or in a previously irradiated area
* Malignant pleural or pericardial effusion.
* Lung tumors with a single additional nodule in the same lobe, same lung or in the contralateral lung, i.e. T3, T4 or M1a lung cancer, in the absence of extrapulmonary involvement.
* Lung involvement in the form of multiple nonsolid or subsolid nodules, in the absence of extrapulmonary metastasis [18]
* History of prior malignant tumour likely to interfere with the protocol treatment or comparisons (excluding H&N primary, radically treated, no recurrence over the last 5 years, non-melanoma skin cancer, in situ cervical cancer, DCIS or LCIS of the breast
* Any relevant co-morbidities that would significantly reduce life expectancy on their own, such as heart failure, advanced COPD, uncontrolled diabetes, end-stage renal disease etc.
* Women who are pregnant or breast feeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | from date of randomization until date of death from any cause up to 60 months
  time interval from randomization until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio V Infante, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona; Michele Milella, PhD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona; Emilio Bria, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Azienda Ospedaliera Universitaria Integrata, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torok JA, Gu L, Tandberg DJ, Wang X, Harpole DH Jr, Kelsey CR, Salama JK. Patterns of Distant Metastases After Surgical Management of Non-Small-cell Lung Cancer. Clin Lung Cancer. 2017 Jan;18(1):e57-e70. doi: 10.1016/j.cllc.2016.06.011. Epub 2016 Jul 5. PMID 27477488
- [Background] Johnson KK, Rosen JE, Salazar MC, Boffa DJ. Outcomes of a Highly Selective Surgical Approach to Oligometastatic Lung Cancer. Ann Thorac Surg. 2016 Oct;102(4):1166-71. doi: 10.1016/j.athoracsur.2016.04.086. Epub 2016 Jun 23. PMID 27344278
- [Background] Ashworth AB, Senan S, Palma DA, Riquet M, Ahn YC, Ricardi U, Congedo MT, Gomez DR, Wright GM, Melloni G, Milano MT, Sole CV, De Pas TM, Carter DL, Warner AJ, Rodrigues GB. An individual patient data metaanalysis of outcomes and prognostic factors after treatment of oligometastatic non-small-cell lung cancer. Clin Lung Cancer. 2014 Sep;15(5):346-55. doi: 10.1016/j.cllc.2014.04.003. Epub 2014 May 15. PMID 24894943
- [Background] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196
- [Background] Iyengar P, Wardak Z, Gerber DE, Tumati V, Ahn C, Hughes RS, Dowell JE, Cheedella N, Nedzi L, Westover KD, Pulipparacharuvil S, Choy H, Timmerman RD. Consolidative Radiotherapy for Limited Metastatic Non-Small-Cell Lung Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2018 Jan 11;4(1):e173501. doi: 10.1001/jamaoncol.2017.3501. Epub 2018 Jan 11. PMID 28973074
- [Background] Yamaguchi M, Edagawa M, Suzuki Y, Toyozawa R, Hirai F, Nosaki K, Seto T, Takenoyama M, Ichinose Y. Pulmonary Resection for Synchronous M1b-cStage IV Non-Small Cell Lung Cancer Patients. Ann Thorac Surg. 2017 May;103(5):1594-1599. doi: 10.1016/j.athoracsur.2016.08.098. Epub 2016 Nov 15. PMID 27863731
- [Background] Detterbeck FC, Franklin WA, Nicholson AG, Girard N, Arenberg DA, Travis WD, Mazzone PJ, Marom EM, Donington JS, Tanoue LT, Rusch VW, Asamura H, Rami-Porta R; IASLC Staging and Prognostic Factors Committee; Advisory Boards; Multiple Pulmonary Sites Workgroup. The IASLC Lung Cancer Staging Project: Background Data and Proposed Criteria to Distinguish Separate Primary Lung Cancers from Metastatic Foci in Patients with Two Lung Tumors in the Forthcoming Eighth Edition of the TNM Classification for Lung Cancer. J Thorac Oncol. 2016 May;11(5):651-665. doi: 10.1016/j.jtho.2016.01.025. Epub 2016 Mar 2. PMID 26944304
- [Background] Conibear J, Chia B, Ngai Y, Bates AT, Counsell N, Patel R, Eaton D, Faivre-Finn C, Fenwick J, Forster M, Hanna GG, Harden S, Mayles P, Moinuddin S, Landau D. Study protocol for the SARON trial: a multicentre, randomised controlled phase III trial comparing the addition of stereotactic ablative radiotherapy and radical radiotherapy with standard chemotherapy alone for oligometastatic non-small cell lung cancer. BMJ Open. 2018 Apr 17;8(4):e020690. doi: 10.1136/bmjopen-2017-020690. PMID 29666135
- [Background] Detterbeck FC, Marom EM, Arenberg DA, Franklin WA, Nicholson AG, Travis WD, Girard N, Mazzone PJ, Donington JS, Tanoue LT, Rusch VW, Asamura H, Rami-Porta R; IASLC Staging and Prognostic Factors Committee; Advisory Boards; Multiple Pulmonary Sites Workgroup. The IASLC Lung Cancer Staging Project: Background Data and Proposals for the Application of TNM Staging Rules to Lung Cancer Presenting as Multiple Nodules with Ground Glass or Lepidic Features or a Pneumonic Type of Involvement in the Forthcoming Eighth Edition of the TNM Classification. J Thorac Oncol. 2016 May;11(5):666-680. doi: 10.1016/j.jtho.2015.12.113. Epub 2016 Mar 3. PMID 26940527
- [Background] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Background] https://evs.nci.nih.gov/ftp1/CTCAE/About.html
- [Background] Seely AJ, Ivanovic J, Threader J, Al-Hussaini A, Al-Shehab D, Ramsay T, Gilbert S, Maziak DE, Shamji FM, Sundaresan RS. Systematic classification of morbidity and mortality after thoracic surgery. Ann Thorac Surg. 2010 Sep;90(3):936-42; discussion 942. doi: 10.1016/j.athoracsur.2010.05.014. PMID 20732521
- [Background] Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. No abstract available. PMID 7713792